CLINICAL TRIAL: NCT06770712
Title: Mirror Therapy as an Adjunct to Bilateral TENS for Improving Upper Extremity Motor Function in Chronic Stroke: A Randomized Controlled Trial
Brief Title: Mirror Therapy Combined With TENS for Motor Recovery in Paretic Upper Limbs of Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeynep ÖZDEMİR, Resident Doctor, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023/273
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-01

CONDITIONS: Hemiplegia
Keywords: Upper extremity motor function; TENS therapy; Mirror therapy; Fugl-Meyer Assessment; Functional improvement
MeSH Terms: conditions — Hemiplegia | interventions — Mirror Movement Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: This study consists of two groups: the Mirror Group and the Control Group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bilateral TENS+ Mirror therapy (Experimental): In addition to conventional treatment, the mirror therapy group received TENS therapy on the finger extensor muscles of both the intact and paretic sides, five times a week for four weeks, with a total of 20 sessions, each lasting 30 minutes. Following TENS therapy, 30 minutes of mirror therapy were administered in each session.
  Interventions: Other: Mirror therapy; Device: Transcutaneous Electrical Nerve Stimulation
- Bilateral TENS (Active Comparator): In addition to conventional treatment, the control group received TENS therapy on the finger extensor muscles of both the intact and paretic sides, five times a week for four weeks, with a total of 20 sessions, each lasting 30 minutes.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Other: Mirror therapy — The patients were asked to sit in front of a table at an appropriate height and rest their arms on the table. A mirror was placed between both arms. The mirror was positioned so that the reflection of the healthy extremity overlapped with the paralytic extremity. In this way, the movements of the healthy upper extremity were viewed through the mirror, creating a visual movement illusion for the hemiplegic upper extremity. During the mirror therapy, exercises including forearm supination-pronation, wrist flexion-extension, finger flexion-extension, finger counting, grasping and releasing a cup, grasping and releasing a ball, and writing with a pen were performed. First, 30 minutes of bilateral TENS therapy were applied, followed by 30 minutes of mirror therapy
  Arms: Bilateral TENS+ Mirror therapy
Device: Transcutaneous Electrical Nerve Stimulation — Received stimulation on the extensor muscles of the hand fingers of both the intact and paretic sides, with a frequency of 100 Hz, pulse width of 200 microseconds, and a biphasic symmetric pulse for 30 minutes. The intensity of the current was adjusted to a level that produced a visible, comfortable muscle contraction. Self-adhesive electrodes, measuring 5x5 cm, were placed on the extensor surface of the forearm, 5 cm distal to the olecranon, parallel to the long axis of the muscle. Electrical stimulation was applied using the Cefar Rehab X2 device (DJO France SAS).

SUMMARY:
The aim of this study is to determine whether mirror therapy, applied in addition to bilateral upper extremity transcutaneous electrical nerve stimulation in patients with chronic stroke, has an additive effect on upper extremity motor recovery

DETAILED DESCRIPTION:
A prospective, single-blind, randomized controlled clinical trial included 30 chronic stroke patients. The patients were assigned to the Mirror group (n=15) and the Control group (n=15) through block randomization.At the end of the three-month follow-up period, 11 patients in the Mirror group and 14 patients in the Control group completed the study. Both groups received conventional rehabilitation therapy for a total of 20 sessions (5 days a week for 4 weeks), along with 30 minutes of transcutaneous electrical nerve stimulation (TENS) applied bilaterally to the finger extensor muscles. In the Mirror group, mirror therapy was additionally administered following the TENS intervention.Upper extremity motor function was assessed by a blinded evaluator using the Fugl-Meyer Assessment for Upper Extremity (FMA-UE) at three time points: baseline, immediately post-treatment (1 month), and at follow-up (2 months after treatment completion).

The effect size (Cohen's d = 0.314) used to calculate the minimum sample size for detecting a significant difference between groups (Bi-TENS + Mirror therapy, Bi-TENS) was obtained from a previous study. (Peiming ve ark. 2021) The sample size was then calculated using the G*Power software version 3.1.9.4 (Franz Faul, University of Kiel, Germany), with an alpha error level of 0.05, a power of 0.95, an inter-correlation of 0.5, and a global non-correlation of 1. The total sample size required for this study was calculated to be 24. Assuming a dropout rate of 20%, the total sample size was determined to be 30.

The normality of the variables was assessed graphically and using the Shapiro-Wilk test. Data that followed a normal distribution were summarized as Mean ± Standard Deviation, while data that did not follow a normal distribution were summarized as Median and the interquartile range (Q1-Q3). Categorical variables were summarized as frequency (percentage). Comparisons of means between groups were performed using the Independent Samples t-test if the data followed a normal distribution, and the Mann-Whitney U test if the data did not follow a normal distribution. For categorical variables, comparisons between groups were made using the Chi-square test or Fisher's Exact test. Intra-group comparisons of means were performed using repeated measures ANOVA. Bonferroni correction was applied for post-hoc pairwise comparisons. A statistical significance level of p < 0.05 was considered. The data were statistically analyzed using the per-protocol approach. Additionally, the intention-to-treat analysis was performed using the Last Observation Carried Forward (LOCF) method. In the LOCF method, missing values are replaced with the last available observation for each participant Statistical analyses and calculations were performed using IBM SPSS Statistics 21.0 (IBM Corp. Released 2012. IBM SPSS Statistics for Windows, Version 21.0. Armonk, NY: IBM Corp.) and MS-Excel 2007.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a history of unilateral stroke
* Cases with a stroke duration of >6 months
* Brunnstrom stage for the upper extremity ≥3
* Brunnstrom stage for the hand ≥4
* Mini-mental test score >21
* Normal vision and hearing functions

Exclusion Criteria:

* Individuals with aphasia
* Individuals with neglect
* Those with a history of traumatic brain injury
* Individuals with uncontrolled cardiovascular disease
* Active inflammatory rheumatological or infectious diseases
* Individuals with significant upper extremity peripheral neuropathy
* Those with severe sensory deficits
* Individuals with severe shoulder, elbow, wrist, or finger severe spasticity(Modified Ashworth Scale score of 4)
* Individuals with a cardiac pacemaker
* Those with lesions on the skin of the upper extremity
* Individuals with skin allergies

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment for Upper Extremity | Change from baseline in the Fugl-Meyer Motor Assessment Scale immediately post-treatment (1 month) and 2 months after treatment completion.
  The Fugl-Meyer Motor Assessment Scale evaluates reflex activity, synergy, and non-synergistic patterns, as well as motor skills and coordination, reflecting the stages of motor development. This assessment consists of a total of 33 items, with each item scored on a 2-point scale. When scoring for the upper extremity, a participant can receive a maximum of 66 points. In the upper extremity assessment, a score of 53-66 points is classified as full capacity, 48-52 points as sufficient capacity, 32-47 points as limited capacity, and 31 points or below as weak capacity.

CONTACTS AND LOCATIONS:
Overall Officials: İlhan KARACAN, Professor Doctor, Study Director — T.C SAĞLIK BİLİMLERİ ÜNİVERSİTESİ İSTANBUL FİZİK TEDAVİ REHABİLİTASYON EĞİTİM VE ARAŞTIRMA HASTANESİ
Locations (1):
- T.C Sağlik Bilimleri Üniversitesi İstanbul Fizik Tedavi Rehabilitasyon Eğitim Ve Araştirma Hastanesi, Istanbul, BAHÇELİEVLER, Turkey (Türkiye)